CLINICAL TRIAL: NCT00017485
Title: A Phase I Study Of Photodynamic Therapy (PDT) For The Treatment Of Basal Cell Carcinoma (BCC): A Drug/Light Dose Finding Study Utilizing 2-(1-HEXYLOXYETHYL)-2-DEVINYL PYROPHEOPHORBIDE-A (HPPH-PHOTOCLOR)
Brief Title: Photodynamic Therapy in Treating Patients With Basal Cell Skin Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Alan Oseroff, MD, Roswell Park Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068696; P30CA016056 (NIH); RPCI-DS-95-34; NCI-G01-1953
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Non-melanomatous Skin Cancer
Keywords: basal cell carcinoma of the skin; recurrent skin cancer
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Neoplasms | interventions — 2-(1-hexyloxyethyl)-2-devinyl pyropheophorbide-a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: HPPH

SUMMARY:
RATIONALE: Photodynamic therapy uses light and drugs that make cancer cells more sensitive to light to kill tumor cells. Photosensitizing drugs such as HPPH are absorbed by cancer cells and, when exposed to light, become active and kill the cancer cells.

PURPOSE: Phase I trial to study the effectiveness of photodynamic therapy with HPPH in treating patients who have basal cell skin cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of HPPH used in photodynamic therapy in patients with basal cell skin cancer.
* Determine the drug dose, light dose, and treatment interval combinations that do not produce excessive toxicity to normal skin but effect tumor response in these patients treated with this regimen.
* Determine the length of time for cutaneous photosensitivity in these patients treated with this regimen.
* Determine the plasma clearance rates for HPPH in these patients.
* Determine the best combination of treatment parameters for a phase II study.

OUTLINE: This is a dose-escalation study.

Patients receive HPPH IV on day 1. Patients undergo phototherapy on days 2-3.

Cohorts of 2-6 patients receive escalating doses of HPPH and phototherapy to determine the minimum erythemal dose (MED). The MED is defined as the dose combination of HPPH and laser light preceding that at which at least 1 patient experiences grade 3 or worse toxicity or at which at least 2 patients experience grade 1 or worse toxicity.

Patients are followed daily for 4 days, at week 1, and at months 1, 3, 6, 12, and 24.

PROJECTED ACCRUAL: A total of 4-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-morpheaform basal cell skin cancer

  * Primary disease OR
  * Recurrent disease after prior therapy (e.g., surgical excision, electrodesiccation, cryosurgery, or radiotherapy)
* At least 4 lesions, no greater than 2 cm in diameter and no greater than 5 mm in depth
* No lesions located on the eyelid, nose, ear, periauricular area, genitals, or digits, or any other lesions thought to be deep and/or aggressive

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 120,000/mm^3

Hepatic:

* PT/PTT no greater than 1.5 times upper limit of normal (ULN)
* Bilirubin no greater than 3.0 mg/dL
* Liver enzymes no greater than 2 times ULN
* No impaired hepatic function

Renal:

* No impaired renal function

Cardiovascular:

* No myocardial infarction within the past 6 months

Other:

* No porphyria
* No known hypersensitivity to porphyrins
* No systemic lupus erythematosus
* No history of positive antinuclear antibody
* No history of degenerative disease of the retina
* No xeroderma pigmentosum
* No pancreatic disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 3 months since prior combination doxorubicin and radiotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* See Chemotherapy

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2000-01; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan R. Oseroff, MD, PhD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States